CLINICAL TRIAL: NCT01309906
Title: A Study to Evaluate the Product Feasibility of a New Silicone Hydrogel Contact Lens
Brief Title: Evaluation of the Feasibility a New Silicone Hydrogel Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 688E
Record Dates: First submitted 2011-03-04; First posted 2011-03-07 (Estimated); Results first posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-09

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Investigational lens (Experimental): Bausch & Lomb investigational silicone hydrogel lens
  Interventions: Device: Investigational lens
- Air Optix Aqua lens (Active Comparator): Ciba Vision Air Optix Aqua contact lens
  Interventions: Device: Air Optix Aqua lens

INTERVENTIONS:
Device: Investigational lens — Bausch & Lomb investigational silicone hydrogel contact lens worn on a daily wear basis for 1 week.
  Arms: Investigational lens
Device: Air Optix Aqua lens — Ciba Visions Air Optix Aqua contact lens, worn on a daily wear basis for 1 week.
  Arms: Air Optix Aqua lens

SUMMARY:
The objective of this study is to determine the clinical feasibility and to evaluate the product performance of an investigational contact lens.

ELIGIBILITY:
Inclusion Criteria:

* Have physiologically normal anterior segments not exhibiting clinically significant biomicroscopy findings.
* Be myopic and require lens correction in each eye.
* Be adapted wearers of soft contact lenses, wear a lens in each eye, and each lens must be of the same manufacture and brand.

Exclusion Criteria:

* Any systemic disease affecting ocular health.
* Using any systemic or topical medications that will affect ocular physiology or lens performance.
* An active ocular disease, any corneal infiltrative response or are using any ocular medications.
* Any "Present" finding during the slit lamp examination that, in the Investigator's judgment, interferes with contact lens wear.
* Allergic to any component in the study care products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2010-12; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tara Vaz, OD, Principal Investigator — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb Incorporated, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 66 participants (132 eyes) were enrolled in the study. One-half were randomized to receive the investigational lens, and the other half were randomized to receive the control lens. After one week of wearing the first lens type, the subjects returned for an exam and crossed over to the second lens type for one week.
Groups:
- Investigational Lens Then Air Optix Aqua Lens: Bausch & Lomb investigational silicone hydrogel lens
  Investigational lens: Bausch & Lomb investigational silicone hydrogel contact lens worn on a daily wear basis for 1 week.
  Ciba Vision Air Optix Aqua contact lens Air Optix Aqua lens: Ciba Visions Air Optix Aqua contact lens, worn on a daily wear basis for 1 week.
- Air Optix Aqua Lens Then Investigational Lens: Ciba Vision Air Optix Aqua contact lens
  Air Optix Aqua lens: Ciba Visions Air Optix Aqua contact lens, worn on a daily wear basis for 1 week.
  Bausch & Lomb investigational silicone hydrogel lens Investigational lens: Bausch & Lomb investigational silicone hydrogel contact lens worn on a daily wear basis for 1 week.
Period: Overall Study
Arm/Group | Investigational Lens Then Air Optix Aqua Lens | Air Optix Aqua Lens Then Investigational Lens
Started | 33 | 33
Completed | 32 | 32
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Overall: All participants received both treatment groups.
Arm/Group | Overall
Number analyzed (Participants) | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.1 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 22

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity
Description: Visual acuity was assessed by distance high contrast logarithm of the minimum angle of resolution (logMAR).
Time Frame: At 1 week follow up
Population: There were 65 subjects (130 eyes) in each group for this outcome measure.
Measure: Least Squares Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Investigational Lens | Air Optix Aqua Lens
Number analyzed (Participants) | 65 | 65
Number analyzed (eyes) | 130 | 130
logMAR | -0.038 (0.088) | -0.040 (0.088)

2. Secondary Outcome: Percentage of Eyes With > Grade 2 Slit Lamp Findings
Description: Graded slit lamp findings for each eye, including epithelial edema, epithelial microcysts, corneal staining, limbal and bulbar injections, upper lid tarsal conjunctival abnormalities, corneal neovascularization, and corneal infiltrates were graded for severity on a scale from 0 (No Finding) to 4 (Severe Finding). The outcome measure is any finding > grade 2, across abnormalities.
Time Frame: At 1 week follow up
Population: There were 65 subjects (130 eyes) in each group for this outcome measure.
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Investigational Lens | Air Optix Aqua Lens
Number analyzed (Participants) | 65 | 65
Number analyzed (eyes) | 130 | 130
eyes | 0 | 0

3. Secondary Outcome: Symptoms and Complaints
Description: At 1-Week Follow-up, subjects were asked to rate 16 common symptoms/complaints on a scale of 0 to 100, with 100 being the most favorable score.
Time Frame: At 1 week follow up
Population: There were 65 subjects (130 eyes) in each group for this outcome measure.
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Investigational Lens | Air Optix Aqua Lens
Number analyzed (Participants) | 65 | 65
Number analyzed (eyes) | 130 | 130
score on a scale
  Burning/stinging upon insertion | 89.7 (16.7) | 90.5 (16.7)
  Comfort upon insertion | 86.6 (18.9) | 86.9 (18.9)
  Overall comfort | 85.7 (18.4) | 87.8 (18.4)
  Comfort at end of day | 80.1 (22.7) | 79.2 (22.7)
  Ease of handling/insertion | 86.3 (17.8) | 91.7 (17.8)
  Ease of handling/removal | 90.7 (13.0) | 93.2 (13.0)
  Dryness | 83.0 (19.8) | 81.8 (19.8)
  Itchiness | 90.2 (16.2) | 90.4 (16.2)
  Redness | 92.1 (11.3) | 93.1 (11.3)
  Vision upon insertion | 88.1 (14.8) | 92.7 (14.8)
  Vision | 88.3 (14.8) | 90.7 (14.8)
  Vision in low light | 86.9 (14.9) | 88.6 (14.9)
  Lens cleanness upon insertion | 91.6 (12.2) | 93.4 (12.2)
  Lens cleanness upon removal | 87.4 (17.6) | 89.5 (17.6)
  Overall impression | 83.9 (19.4) | 84.5 (19.4)
  Lens cleanness | 87.9 (17.0) | 89.6 (17.0)

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: Adverse events were not coded. Therefore source vocabulary is not applicable.
Arm/Group | Investigational Lens | Air Optix Aqua Lens
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/66
Other Adverse Events (participants affected / at risk) | 0/66 | 0/66

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.